CLINICAL TRIAL: NCT07279233
Title: A Phase 1, Open-Label Study to Assess the Enzyme Inducing Effects of Carbamazepine on the Pharmacokinetics of Mirdametinib and Its Metabolites in Healthy Participants
Brief Title: To Assess the Enzyme Inducing Effects of Carbamazepine on the PK of Mirdametinib in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEK-NF1-105
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Volunteer
Keywords: Drug interaction, mirdametinib, carbamazepine
MeSH Terms: interventions — mirdametinib; Carbamazepine

STUDY DESIGN:
Intervention Model Description: Fixed-sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 Mirdametinib (Active Comparator): Mirdametinib 6-mg single dose given orally alone on Day 1 as three 2-mg capsules following a 10-hour fast.
  Interventions: Drug: Mirdametinib
- Period 2 Mirdametinib and carbamazepine (Experimental): Mirdametinib 6-mg single dose given orally on Day 22 in Period 2 as three 2-mg capsules following a 10-hour fast in combination with carbamazepine tablets that are administered orally according to the following schedule:
  * Days 8 and 9: 100 mg BID with meals
  * Days 10 and 11: 200 mg BID with meals
  * Days 12 through 21: 300 mg BID with meals
  * Day 22: 300 mg AM fasted, with mirdametinib, and 300 mg PM with meal
  * Days 23 through 28: 300 mg BID with meals
  * Days 29 through 30: no doses (observation only)
  Interventions: Drug: Mirdametinib and Carbamazepine

INTERVENTIONS:
Drug: Mirdametinib — 6-mg single dose given orally on Day 1
  Arms: Period 1 Mirdametinib
Drug: Mirdametinib and Carbamazepine — Drug: Mirdametinib 6-mg single dose given orally on Day 22. Drug: Carbamazepine Carbamazepine extended-release (ER) (Carbamazepine ER will be given orally twice daily for 21 days with a titration schedule [100 mg BID for 2 days, 200 mg BID for 2 days, and then 300 mg BID]).
  Arms: Period 2 Mirdametinib and carbamazepine

SUMMARY:
The purpose of this study is to determine the effect of carbamazepine on the blood levels of mirdametinib and how long it takes the body to eliminate mirdametinib when both drugs are administered orally in healthy participants. The study may last up to approximately 64 days for each participant.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, fixed-sequence, 2-period clinical study in healthy participants. Approximately 36 participants will be enrolled in the study to achieve 25 evaluable participants.

Healthy male and/or female participants, aged 18 to 65 years (inclusive), not of Asian descent, with body mass index (BMI) between 18 and 32 kg/m², and who are medically healthy with no clinically significant abnormalities.

The study consists of screening (28 days), 2 study periods, and a 7-day follow-up.

Mirdametinib will be given as a single 6-mg dose on 2 separate occasions: once on Day 1 and once on Day 22. Carbamazepine ER will be given twice daily for 21 days beginning on Day 8.

On Day 1 of Period 1, participants will receive a 6-mg single oral dose of mirdametinib followed by PK sampling for 168 hours (Day 8). In Period 2, participants will receive carbamazepine extended-release (ER) twice daily for 21 days with a titration schedule (100 mg twice daily [BID] for 2 days, 200 mg BID for 2 days, and 300 mg BID for the remaining days). On Day 22, participants will receive a 6-mg single dose of mirdametinib with the morning dose of carbamazepine ER, followed by PK sampling for 168 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must sign the informed consent form (ICF) prior to any study-related procedures being performed.
2. Participant is male or female and between 18 and 65 years of age (inclusive) at the time of informed consent.
3. Participant has a body mass index (BMI) ≥18 and ≤32 kg/m² (inclusive) at Screening and Day -1.
4. Participant is in good health in the judgment of the investigator on the basis of a medical evaluation performed at Screening, Day -1, and predose on Day 1, and the results of clinical chemistry, hematology, coagulation, and urinalysis tests carried out at Screening and Day -1. Clinical laboratory test results within normal reference range for the population or investigative site, or results within acceptable deviations that are judged to be not clinically significant by the investigator.

   Note: Laboratory values that are out-of-range may be confirmed by a single repeat per investigator discretion.
5. Participant has normal or mildly impaired renal function as estimated by the Chronic Kidney Disease Epidemiology Collaboration formula (i.e., ≥60 mL/min).
6. Participant has sufficiently good venous access in at least 1 arm to confidently enable serial blood sampling.
7. Male participants who agree to the following during study and for at least 90 days after the last dose of study medication:

   1. Refrain from donating or preserving sperm, PLUS either
   2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR
   3. Must agree to use a male condom when having sexual intercourse with women of childbearing potential (WOCBP). An additional form of contraception should also be used by the female partner if she is of childbearing potential.
8. Female participants that are not pregnant or breastfeeding, and for whom one of the following conditions applies:

   1. Is a woman of non-childbearing potential.
   2. Is a WOCBP and agrees to use an acceptable contraceptive method from the time of signed informed consent and for at least 6 weeks after the last dose of study medication; AND
9. All female participants must have a negative serum pregnancy test at Screening and CRU admission (Day -1)

Exclusion Criteria:

* Participant has clinically significant infections (e.g., coronavirus disease 2019 [COVID-19] or influenza) within 90 days prior to Day 1, as judged by the investigator, or evidence of any infection within 14 days prior to Day 1. If a participant tests positive (reactive) for Hepatitis B, Hepatitis C, or HIV at Screening, they are not eligible for participation in the study.

  2. Participant has a history of any neurological conditions including movement disorders and seizures.

  3. Participant has a history of stomach or GI surgery or resection that would potentially alter absorption, metabolism, and/or excretion of PO administered drugs (exceptions include participants who underwent appendectomy or any type of hernia repair).

  4. Participant has a history of pre-existing condition interfering with normal GI anatomy or motility and potentially alter the absorption, metabolism, and/or excretion of orally administered drugs.

  5. Participants with a history of inflammatory bowel disease, peptic ulceration, or pancreatitis within 180 days prior to Day 1.

  6. Participant has a history of cancer, except if judged to be in full remission for at least 5 years at the time of informed consent (except basal cell skin cancer, resected prostate cancer with an undetectable Prostate-Specific Antigen test (PSA), or squamous cell skin cancer with history of curative treatment and no recurrence for at least 3 years prior to Screening), as judged by the investigator.

  7. Participant has an acute illness with symptoms or treatment that has started or persisted within 14 days prior to Day 1 unless mild in severity and enrollment is approved by both the investigator and the sponsor's medical monitor.

  8. Participant has any evidence of glaucoma or retinal vein occlusion, visual blurring or uncorrected vision issues, or intraocular pressure (IOP) >21 mmHg on Day -1.

  9. Participant has cardiovascular abnormalities including:
  1. History of postural hypotension, unexplained syncope, or abnormal autonomic tone
  2. Blood pressure <90/50 mmHg or >140/90 mmHg after 5 minutes of rest
  3. Heart rate <45 or >100 bpm after 5 minutes of rest
  4. Abnormal QT interval corrected by Fridericia's formula (QTcF) interval (≥450 msec) or ECG abnormalities interfering with QT/QTc interpretation
  5. Risk factors for torsades de pointes
  6. Ejection fraction <55% 10. Participant has an acute illness, significant infection, or incomplete bladder emptying (voiding >2 times/night).

     11. Participant has any clinically significant abnormality in hematology parameters at Screening or Day -1 as determined by the investigator.

  <!-- -->

  1. Participant has a hemoglobin < 11.0 g/dL for female participants or < 12.5 g/dL for male participants.
  2. Participant has a hematocrit < the lower limit of normal.
  3. Participant has a white blood cell count < the lower limit of normal.
  4. Participant has a platelet count < the lower limit of normal. 12. Participant has a history or evidence of any hematological disorder such as anemia, leukopenia, thrombocytopenia, or bleeding disorder.

     13. Participant has any known or suspected hereditary blood disorder (e.g., sickle cell, or thalassemia).

     14. Participant has alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or total bilirubin levels >1.5× the upper limit of normal at Screening or Day -1.

     15. Participant has substance use concerns:

  <!-- -->

  1. Positive alcohol, cotinine, or drug screen test
  2. Alcohol intake >3 units/day or >14 units/week in past 6 months
  3. Excessive caffeine consumption (>400 mg/day)
  4. Tobacco or nicotine use within 3 months of Screening
  5. Unwillingness to avoid xanthine-containing products 72 hours before dosing 16. Participant has taken, received, or consumed:

  <!-- -->

  1. Any prescription medications, over-the-counter medications, supplements, or herbal products within 28 days or 5 half-lives if known (whichever is longer)
  2. Vaccines within 14 days prior to Day 1; live vaccines within 28 days prior to Day 1.c. Investigational products within 28 days or 5 half-lives, or >3 new investigational entities within 12 months

  d. Red wine, any fruit juices (including, but not limited to, grapefruit, grapefruit juice, pomelos, or other exotic citrus fruits, or grapefruit hybrids), or any nutrients known to modulate drug metabolizing enzyme/transporters activity (including, but not limited to, cranberries or star fruits) within 72 hours of Day -1 17. Participant has donated blood (>450 mL) within 60 days, donated plasma within 7 days, or received blood products within 60 days.

  18. Participant is unwilling to avoid strenuous activity, sunbathing, or contact sports during the study.

  19. Participant has a history of known prior major depression. 20. Participant has a significant risk of committing suicide based on medical history in the opinion of the investigator; or an answer of "Yes" to questions #4 or #5 of the Columbia-Suicide Severity Scale (C-SSRS; [Posner 2011]).

  21. Participant has specific contraindications to the study medications:

  a. Known hypersensitivity to carbamazepine, mirdametinib, or related compounds b. Participant is Asian or has one or more Asian parents or grandparents c. History of anaphylaxis d. History of severe cutaneous adverse reactions (such as Stevens-Johnson Syndrome, toxic epidermal necrolysis, or Drug Reaction with Eosinophilia and Systemic Symptoms).

  22. Participant is deemed unsuitable for this study in the opinion of the investigator for any additional reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The geometric mean ratio of mirdametinib plasma area under the concentration-time curve from dosing extrapolated to infinity (AUCinf) of Mirdametinib | Day 1 to Day 29
The geometric mean ratio area under the concentration-time curve from dosing to time of last quantifiable concentration (AUClast) of Mirdametinib | Day 1 to Day 29
The geometric mean ratio of maximum observed concentration (Cmax) of Mirdametinib | Day 1 to Day 22

SECONDARY OUTCOMES:
Number of participants who Experience an Adverse Event | Up to a maximum of 36 days
AUCinf of Metabolites M15, M22, and M30 | Day 1 to Day 29
AUClast of Metabolites M15, M22, and M30 | Day 1 to Day 29
Cmax of Metabolites M15, M22, and M30 | Day 1 to Day 22
Time of maximum observed concentration (Tmax) of Mirdametinib and Metabolites M15, M22, and M30 | Day 1 to Day 22
Apparent terminal elimination half-life (t1/2) of Mirdametinib and Metabolites M15, M22, and M30 | Day 1 to Day 29
Apparent clearance (CL/F) of Mirdametinib and Metabolites M15, M22, and M30 | Day 1 to Day 29
Apparent volume of distribution (Vd/F) of Mirdametinib and Metabolites M15, M22, and M30 | Day 1 to Day 29
Metabolite to parent molar ratio AUCinf (MRAUCinf) | Day 1 to Day 29
  (AUCinf, metabolite/MWmetabolite)/(AUCinf, parent/MWparent)
Metabolite to parent molar ratio AUClast (MRAUClast), | Day 1 to Day 29
  (AUClast, metabolite/MWmetabolite)/(AUClast, parent/MWparent)
Metabolite to parent molar ratio Cmax (MRCmax) | Day 1 to Day 22
  (Cmax, metabolite/MWmetabolite)/(Cmax, parent/MWparent)

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent participant-level data from completed clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.